CLINICAL TRIAL: NCT02388919
Title: A Registered Randomized, Double-Blind, Placebo-Controlled (2:1), Multi-Centered Clinical Trial of Anlotinib as a Treatment for Advanced Non-Small Cell Lung Cancer
Brief Title: Study of Anlotinib in Patients With Advanced Non-small Cell Lung Cancer（ALTER0303）
Acronym: ALTER0303
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-03-IIB
Record Dates: First submitted 2015-02-25; First posted 2015-03-17 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: anlotinib; Cancer; NSCLC; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anlotinib (Experimental): Anlotinib p.o, qd and it should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo p.o, qd and it should be continued until disease progress or patients withdraw consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Basic dosage, take once when limosis in the morning. If patients cannot suffer from AEs, they can get declined dosage.
  Other Names: AL3818
  Arms: Anlotinib
Drug: Placebo — Basic dosage, take once when limosis in the morning.
  Arms: Placebo

SUMMARY:
Evaluate the efficacy and safety of Anlotinib as the 3-line treatment of patients with advanced non-small lung cancer, with placebo control.

DETAILED DESCRIPTION:
Anlotinib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β c-Kit and MET.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Diagnosed with advanced NSCLC (phase IIIB/IV) through pathology, with measurable nidus(using RECIST 1.1)
3. at least two systematic chemotherapy with upwards of 3-line treatments or cannot suffer
4. Patients must provide detectable specimen (from tumor tissue or hydrothorax) before participating, who negative in EGFR&ALK can participate or who positive in EGFR&ALK, have or have not drug tolerance after the treatment with relative targeted drugs
5. ECOG PS：0-1,Expected Survival Time: Over 3 months
6. main organs function is normal
7. The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it

Exclusion Criteria:

1. have used Anlotinib before
2. Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer)
3. examined as positive in EGFR&ALK mutation detection and never take the treatment of TKIs
4. central lung squamous carcinoma along with cavum, or non-small cell lung cancer along with hemoptysis (>50ml/day)
5. other kinds of malignancies within 5 years or for now
6. plan to take systemic anti-tumor therapy within 4 weeks before grouping or during the medicine-taking period of this research, including Cytotoxic Therapy, Signal Transduction Inhibitor, and Immunotherapy (or who use Mitomycin C within 6 weeks before taking the treatment with experimental drug); The patients who have already taken Extended Field Radiotherapy (EF-RT) within 4 weeks before grouping or Limited Field Radiotherapy with proposed assessment of nidus within 2 weeks before grouping
7. have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
8. with kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus)
9. pleural effusion or ascites, resulting in respiratory syndrome (≥CTC AE level 2)
10. symptoms of brain metastases cannot be controlled and treated within less than 2 months
11. get any severe diseases or the ones that cannot be controlled
12. take major surgical treatments, open biopsy, or get overt traumatic injury within 28 days before grouping
13. have any habitus or medical history of hemorrhage, however severe it is; the patients who have non healing wounds, ulcer or fracture after any events with hemorrhage or bleeding (≥CTCAE level 3)
14. get arterial/venous thrombosis within 6 months, such as cerebrovascular accidents (including temporary ischemic stoke), deevenous thrombosis, and pulmonary embolism
15. ever abuse psychiatric drugs and cannot abstain or who are diagnosed with mental disorder
16. have participated in other clinical trials of anti-tumor medicine within 4 weeks
17. diagnosed with disease which will severely endanger the security of patients or influence the completion of this research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)

SECONDARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death(up to 24 months)
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until 30 day safety follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, professor, Study Director — Chest hospital affiliated to Shanghai jiaotong university; Kai Lee, professor, Study Director — Tianjin Medical University Cancer Hospital
Locations (40):
- China (40):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Capital Medical University, Beijing Chest Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, Chongqing, Chongqing Municipality
  - Fujian Province Tumor Hospital, Fuzhou, Fujian
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Gansu Provincial People 's Hospital, Lanzhou, Gansu
  - Lanzhou Military General Hospital, Lanzhou, Gansu
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin medical university affiliated tumor hospita, Harbin, Heilongjiang
  - Henan Province Tumor Hospital, Luoyan, Henan
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Lianyungang First People 's Hospital, Lianyungang, Jiangsu
  - Xuzhou Medical College Hospital, Xuzhou, Jiangsu
  - Jiangxi Province Tumor Hospital, Nanchang, Jiangxi
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - Liaoning Provincial Tumor Hospital, Shenyang, Liaoning
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Shandong Province Tumor Hospital, Jinan, Shandong
  - Linyi City Tumor Hospita, Linyi, Shandong
  - Chest hospital affiliated to Shanghai jiaotong university, Shanghai, Shanghai Municipality
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Xinhua hospital affiliated to Shanghai jiaotong university, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - Tang Du Hospital, Xian, Shanxi
  - West China Hospital , Sichuan University, Chengdu, Sichuan
  - Sichuan Cancer Hospital, Chongqing, Sichuan
  - 20th Floor, Block C, Lake Road, Hexi District, Tianjin Medical University Cancer Institute and Hospital ., Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Yunnan Province Tumor Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Province Tumor Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qin T, Liu Z, Wang J, Xia J, Liu S, Jia Y, Liu H, Li K. Anlotinib suppresses lymphangiogenesis and lymphatic metastasis in lung adenocarcinoma through a process potentially involving VEGFR-3 signaling. Cancer Biol Med. 2020 Aug 15;17(3):753-767. doi: 10.20892/j.issn.2095-3941.2020.0024. PMID 32944404
- [Derived] Jiang S, Liang H, Liu Z, Zhao S, Liu J, Xie Z, Wang W, Zhang Y, Han B, He J, Liang W. The Impact of Anlotinib on Brain Metastases of Non-Small Cell Lung Cancer: Post Hoc Analysis of a Phase III Randomized Control Trial (ALTER0303). Oncologist. 2020 May;25(5):e870-e874. doi: 10.1634/theoncologist.2019-0838. Epub 2020 Feb 20. PMID 32077550
- [Derived] Zhang PL, Liu ZJ. Esophago-tracheobronchial fistula following treatment of anlotinib in advanced squamous cell lung cancer: Two case reports. Medicine (Baltimore). 2019 Nov;98(44):e17700. doi: 10.1097/MD.0000000000017700. PMID 31689797
- [Derived] Si XY, Wang HP, Zhang XT, Wang MZ, Zhang L. [Efficacy and safety of anlotinib in 16 patients with advanced non-small cell lung cancer]. Zhonghua Nei Ke Za Zhi. 2018 Nov 1;57(11):830-834. doi: 10.3760/cma.j.issn.0578-1426.2018.11.007. Chinese. PMID 30392239
- [Derived] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Derived] Si X, Zhang L, Wang H, Zhang X, Wang M, Han B, Li K, Wang Q, Shi J, Wang Z, Cheng Y, He J, Shi Y, Chen W, Wang X, Luo Y, Nan K, Jin F, Li B, Chen Y, Zhou J, Wang D. Quality of life results from a randomized, double-blinded, placebo-controlled, multi-center phase III trial of anlotinib in patients with advanced non-small cell lung cancer. Lung Cancer. 2018 Aug;122:32-37. doi: 10.1016/j.lungcan.2018.05.013. Epub 2018 May 18. PMID 30032842
- See also: official website — http://www.cttq.com/